CLINICAL TRIAL: NCT00536211
Title: Physical Inactivity and Insulin Resistance in Skeletal Muscle.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol not approved by VA R&D
Sponsor: University of Kansas Medical Center (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1095378
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2015-08

CONDITIONS: Metabolic Syndrome X; Insulin Resistance; Hypertension; Hypercholesterolemia; Obesity
Keywords: Exercise; Physical Activity; Metformin; Hyperinsulinemic-Euglycemic Clamp; Muscle Biopsy; Fatty Acid Oxidation; Peroxisome proliferator-activated receptor gamma; Detraining; Inactivity; Skeletal muscle
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Hypertension; Hypercholesterolemia; Obesity; Motor Activity; Sedentary Behavior | interventions — Exercise; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise
  Interventions: Behavioral: Exercise
- 2 (Active Comparator): Metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Behavioral: Exercise — Exercise training will consist of walking and/or jogging on a treadmill 5 out of 7 d each week at ~60% of each subject's predetermined VO2max (75% maximal heart rate as monitored by heart rate monitors), 45 min/session, for 12 weeks. The exercise training will follow a three-stage progression: 1. wk 1 = 30 min, 3 d/wk, 60% VO2max; 2. wk 2 = 30 min, 5 d/wk, 60% VO2max; and 3. wk 3-12 = 45 min, 5 d/wk, 60% VO2max.
  Arms: 1
Drug: Metformin — oral tablet, 1000 mg daily for 17 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine how a decline in physical activity acutely leads to a decrease in insulin sensitivity in skeletal muscle. The hypothesis is that the loss of insulin sensitivity following physical inactivity is caused by a rapid reduction in skeletal muscle mitochondrial oxidative capacity.

DETAILED DESCRIPTION:
In this project we will study two diverse groups of subjects. Group 1 will be subjects who are sedentary, insulin resistant, and have the Metabolic Syndrome. These subjects will be tested for insulin sensitivity at the whole body level, and for key changes in skeletal muscle metabolism at baseline, following 12 weeks of exercise training, and during an acute (1-3 days) period of time following the cessation of exercise training. The design allows us to study the effects of exercise on improving insulin sensitivity and make direct comparisons to a period when insulin sensitivity quickly decreases because of the removal of exercise training. Metformin is a drug commonly prescribed to control insulin resistance and type 2 diabetes. Metformin is thought to have exercise like effects on muscle metabolism and is known to activate a molecule that is de-activated during inactivity. Thus, half of the Metabolic Syndrome subjects will cease exercise training with no treatment while another half will quite exercise training while taking the drug Metformin.

Group 2 subjects will be highly trained endurance athletes. Endurance athletes display high levels of insulin sensitivity that can drop in the hours and days following the cessation of exercise. Thus we will take the same measurements in endurance athletes at baseline during their normal training regimen and in the acute (1-3 days) period following the cessation of exercise training. Again, half of the subjects will be take Metformin during the cessation of exercise in the same fashion as done in group 1.

Studies in both groups seek to determine the event(s) which cause insulin resistance in skeletal muscle following a decrease in physical activity levels. Comparisons between healthy, active individuals and sedentary Metabolic Syndrome subjects may provide additional information about the underlying events that cause insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Selection of inclusion for Metabolic Syndrome Subjects :

Sedentary metabolic syndrome subjects will be 20-55 y of age, overweight to Class I or II obese (BMI 25-39 kg/m2) men and women, who have a fasting glucose of 100 to 125 mg/dl, and at least 2 of 4 other characteristics of the metabolic syndrome which are the following: waist circumference greater than 102 cm in men and 88 cm in women, serum triglyceride concentration greater than 150 mg/dl, HDL-C concentration greater than 40 mg/dl in men and 50 mg/dl in women, and blood pressure greater than 130/85 mmHG.

Selection for inclusion for Endurance Athlete Subjects:

Subjects who report training (running and/or biking) greater than 30 min a day, 4 days a week for at least 1 year will be included. Final inclusion criteria will be a VO2max of greater than 55 ml/kg/min.

To take part in the study, Women must currently be taking birth control or be postmenopausal.

Exclusion Criteria:

* Subjects will be excluded from the study if they have or are:

Diagnosed cardiovascular disease or diabetes or disease symptoms that could alter their ability to perform exercise, fasting blood glucose of greater than 126 mg/dl, smokers, taking any medications or supplements (e.g., statins, fibrates, metformin, thiazolidinediones, anti-hypertensives (ACE-inhibitors and angiotensin blockers) which could affect blood lipids or insulin sensitivity.

Women who are pregnant or plan to become pregnant during the duration of the study For the Metabolic Syndrome subjects only individuals exercising regularly (more than one 30 min session per week) or have a physically active lifestyle (>8,000 daily steps as measured by a pedometer) will be excluded.

Individuals with an orthopedic limitations for walking. Allergies to drugs used in the study. Past or current liver and/or kidney problems of any nature.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity; following 12 weeks of exercise training and 1 and 3 days of detraining and + or - Metformin. | 12 weeks and 3 days

SECONDARY OUTCOMES:
PGC-1 alpha transcription and mitochondrial fatty acid oxidation and enzyme activity in skeletal muscle; following 12 weeks of exercise training and 1, 2, and 3 days of detraining and + or - Metformin. | 12 weeks and 3 days

CONTACTS AND LOCATIONS:
Overall Officials: John P Thyfault, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Harry S. Truman Memorial Veterans' Hospital, Columbia, Missouri, United States

REFERENCES:
- [Background] Shulman GI. Cellular mechanisms of insulin resistance. J Clin Invest. 2000 Jul;106(2):171-6. doi: 10.1172/JCI10583. No abstract available. PMID 10903330
- [Background] Haapanen N, Miilunpalo S, Pasanen M, Oja P, Vuori I. Agreement between questionnaire data and medical records of chronic diseases in middle-aged and elderly Finnish men and women. Am J Epidemiol. 1997 Apr 15;145(8):762-9. doi: 10.1093/aje/145.8.762. PMID 9126003
- [Background] Koves TR, Li P, An J, Akimoto T, Slentz D, Ilkayeva O, Dohm GL, Yan Z, Newgard CB, Muoio DM. Peroxisome proliferator-activated receptor-gamma co-activator 1alpha-mediated metabolic remodeling of skeletal myocytes mimics exercise training and reverses lipid-induced mitochondrial inefficiency. J Biol Chem. 2005 Sep 30;280(39):33588-98. doi: 10.1074/jbc.M507621200. Epub 2005 Aug 3. PMID 16079133
- [Background] Russell AP, Feilchenfeldt J, Schreiber S, Praz M, Crettenand A, Gobelet C, Meier CA, Bell DR, Kralli A, Giacobino JP, Deriaz O. Endurance training in humans leads to fiber type-specific increases in levels of peroxisome proliferator-activated receptor-gamma coactivator-1 and peroxisome proliferator-activated receptor-alpha in skeletal muscle. Diabetes. 2003 Dec;52(12):2874-81. doi: 10.2337/diabetes.52.12.2874. PMID 14633846
- [Background] Suwa M, Egashira T, Nakano H, Sasaki H, Kumagai S. Metformin increases the PGC-1alpha protein and oxidative enzyme activities possibly via AMPK phosphorylation in skeletal muscle in vivo. J Appl Physiol (1985). 2006 Dec;101(6):1685-92. doi: 10.1152/japplphysiol.00255.2006. Epub 2006 Aug 10. PMID 16902066
- [Background] Kawate R, Yamakido M, Nishimoto Y, Bennett PH, Hamman RF, Knowler WC. Diabetes mellitus and its vascular complications in Japanese migrants on the Island of Hawaii. Diabetes Care. 1979 Mar-Apr;2(2):161-70. doi: 10.2337/diacare.2.2.161. PMID 520120